CLINICAL TRIAL: NCT00002376
Title: A Randomized Controlled Clinical Study to Determine If the Addition of HIV RNA Viral Load Is an Effective Tool in Determining Treatment Regimens for HIV-Infected Patients
Brief Title: The Effectiveness of HIV RNA Viral Load Testing in Determining Treatment Type in HIV-Infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 246F; MK-0639; 056-00
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-06

CONDITIONS: HIV Infections
Keywords: HIV-1; CD4 Lymphocyte Count; RNA, Viral; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Lamivudine; Stavudine; Zidovudine; Didanosine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
To evaluate, in HIV-infected patients whose baseline CD4 count is 300 to 750 cells/mm3, whether an antiretroviral treatment regimen based upon clinical evaluation and CD4 counts plus HIV RNA viral load is more effective than a treatment regimen based upon clinical evaluation and CD4 counts without the use of HIV RNA viral load information. To assess relative utility of viral load testing in determining therapeutic choice by the surrogate marker of CD4 cell counts after 48 weeks of therapy.

It is hypothesized that among HIV-infected patients whose baseline CD4 count is in the range of 300 to 750 cells/mm3, those patients who incorporate initial and periodic viral RNA measurements in their therapeutic decisions will have higher CD4 counts after 48 weeks than patients whose therapeutic decisions do not incorporate initial and periodic viral RNA measurements.

DETAILED DESCRIPTION:
It is hypothesized that among HIV-infected patients whose baseline CD4 count is in the range of 300 to 750 cells/mm3, those patients who incorporate initial and periodic viral RNA measurements in their therapeutic decisions will have higher CD4 counts after 48 weeks than patients whose therapeutic decisions do not incorporate initial and periodic viral RNA measurements.

Approximately 540 patients are stratified on the basis of baseline CD4 counts and are randomized to one of two treatment groups: 1. viral RNA treatment group or 2. non viral RNA treatment group. Treatment modification is based upon CD4 count, viral RNA levels (group 1 only) and clinical evaluation. Patients receive one of the three antiretroviral treatments:

1. No antiretroviral therapy.
2. Double reverse transcriptase inhibitor (RTI) therapy consisting of any two therapy combinations of: didanosine (ddI), lamivudine (3TC), stavudine (d4T) or zidovudine (ZDV), based upon the treating physician's judgment. The preferred combinations are ZDV + 3TC, d4T + 3TC or ddI + d4T.
3. Triple antiretroviral therapy consisting of double antiretroviral therapy plus indinavir.

Treatment decisions are based upon a standardized algorithm as follows:

CD4 count 500-750 + viral RNA < 10,000:

Group 1: No retroviral therapy. Group 2: No retroviral therapy.

CD4 count 500-750 + viral RNA >= 10,000:

Group 1: Triple therapy. Group 2: No retroviral therapy.

CD4 count 300-499 + viral RNA < 10,000:

Group 1: Double retroviral therapy. Group 2: Double retroviral therapy.

CD4 count 300-499 + viral RNA >= 10,000:

Group 1: Triple therapy. Group 2: Double retroviral therapy.

CD4 count 200-299 + viral RNA < 10,000:

Group 1: Maintain same retroviral therapy unless: there is a CD4 count decrease of 25-49% within 24 weeks of the count falling in the range of 300-499 in which case both retroviral therapies are changed, there is a CD4 count decrease of >= 50% within the 48 weeks of therapy from the time the CD4 count fell within the range of 300-499 in which case triple therapy is initiated, or there is an AIDS-defining illness in which case triple therapy is initiated.

Group 2: Same as Group 1.

CD4 count 200-299 + viral RNA >= 10,000:

Group 1: Triple therapy. Group 2: Maintain same retroviral therapy unless: there is a CD4 count decrease of 25-49% within 24 weeks of the count falling in the range of 300-499 in which case both retroviral therapies are changed, there is a CD4 count decrease of >= 50% within the 48 weeks of therapy from the time the CD4 count fell within the range of 300-499 in which case triple therapy is initiated, or there is an AIDS-defining illness in which case triple therapy is initiated.

CD4 count < 200:

Group 1: Triple therapy. Group 2: Triple therapy.

ELIGIBILITY:
Inclusion Criteria

Patients must have the following:

CD4 count >= 300 and <= 750 cells/mm3.

Exclusion Criteria

Prior Medication:

Excluded:

Prior protease inhibitor therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Foundation Hospital, San Francisco, California, United States